CLINICAL TRIAL: NCT03742726
Title: Study Assessing the Safety and Performance of Smart Matrix® Dermal Replacement Scaffold in the Treatment of Full-Thickness Wounds Arising From Surgical Excision of Basal Cell or Squamous Cell Carcinomas in Male and Female Adult Patients
Brief Title: Study Assessing the Safety and Performance of Smart Matrix®
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Smart Matrix Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SML002/18
Record Dates: First submitted 2018-10-23; First posted 2018-11-15 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Smart Matrix scaffold (Experimental): Smart Matrix dermal replacement scaffold
  Interventions: Device: Smart Matrix scaffold

INTERVENTIONS:
Device: Smart Matrix scaffold — Smart Matrix dermal replacement scaffold

SUMMARY:
Smart Matrix is a sterile, single layer dermal replacement scaffold. The scaffold consists of a porous matrix of cross-linked human fibrin plus alginate that has been designed and optimised to facilitate wound closure and healing through cellular invasion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 years and 90 years of age, inclusive
* Suspected or histologically proven BCC or SCC, where treatment with a skin graft would be considered following excision of the lesion
* Expected wound following excision surgery between 2 cm and 5 cm in diameter, inclusive
* Negative urine or serum pregnancy test in females of childbearing potential who do not plan to become pregnant during the study
* Able and willing to comply with the protocol and necessary wound care/follow-up
* Patient or legally authorised representative (LAR) able to comprehend and sign informed consent prior to enrolment in the study

Exclusion Criteria:

* Aged <18 years or >90 years of age
* Body mass index >=35 kg/m2
* Patients who are pregnant or breastfeeding females, or female patients who plan to become pregnant during the study
* Patients with Stage 3 or higher BCC or SCC
* Skin lesion of a size that will result in an expected post-surgical wound >5 cm in diameter
* Lesion located over a joint
* Lesion located in an area in which scarring is already present
* Lesion located on the face
* Patients with a chronically inflammatory dermatological condition
* History of smoking within 1 year prior to Screening
* Use of any nicotine-containing product during the study, from Screening and through the last follow-up visit
* Patients with Type 1 diabetes mellitus, newly diagnosed diabetes mellitus (within 3 months prior to Screening), or poorly controlled Type 2 diabetes mellitus
* Diagnosis of peripheral vascular disease or venous stasis in proximity to the lesion to be treated
* Presence of significant immunodeficiency or an immunocompromised condition
* Patients who are currently receiving systemic steroid medications or other medications that might impede wound healing
* Patients on anti-coagulants
* Known history of human immunodeficiency virus infection, Hepatitis B, Hepatitis C, or human papillomavirus
* Known coagulopathy (either acquired or congenital) but not including patients on aspirin or other anti-platelet therapy
* Patients who have received radiotherapy treatment to the area to be treated with Smart Matrix
* Patients who have acute or active Charcot's disease or a significant neuropathic disease
* Patients who have suspected signs of systemic or local infection, as determined by the Investigator based on clinical parameters
* History of hypersensitivity or allergic reaction to any of the constituents of Smart Matrix
* History of hypersensitivity or allergic reaction to unknown allergens
* Patients who have been treated with tissue engineered skin or a biological therapy within 30 days (or as described on labelling) of Screening
* Patients who, in the opinion of the Investigator, have co-morbidities and/or an underlying condition that would impact wound healing
* Participation in a clinical study involving an investigational medication or investigational device within the last 30 days or 5 half-lives
* Unwilling or unable, in the opinion of the Investigator, to comply with the protocol
* Unwilling or unable to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of infection and device-related adverse events | 24 weeks
  Safety

SECONDARY OUTCOMES:
Complete wound healing | 24 weeks, 52 weeks
  Measurement of time to >95% re-epithelisiation of wound
Cosmesis | 24 weeks, 52 weeks
  Assessment of scar formation and development using the Patient and Observer Scar Assessment Scale (POSAS)
Cosmesis | 24 weeks, 52 weeks
  Assessment of scar formation and development using the Vancouver Scar Scale (VSS)
Pain at dressing change | 24 weeks, 52 weeks
  Pain at dressing change assessed using a 10 cm VAS
Dressing change | 24 weeks, 52 weeks
  Number of dressing changes will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Baljit Dheansa, MBBS FRCS, Principal Investigator — Queen Victoria Hospital
Locations (4):
- United Kingdom (4):
  - Poole General Hospital, Poole, Dorset
  - Broomfield Hospital, Chelmsford, Essex
  - Wythenshawe Hospital, Manchester University NHS Foundation Trust, Manchester, Greater Manchester
  - The Queen Victoria Hospital NHS Foundation Trust, East Grinstead, West Sussex